CLINICAL TRIAL: NCT05510362
Title: Management and Short Term Outcome of Traumatic Wounds in the Emergency Department
Acronym: SUTURES
Status: Recruiting | Type: Observational
Sponsor: University of Monastir (Other)
Responsible Party: Principal Investigator, Pr. Semir Nouira, professor, University of Monastir
Other Study IDs: SUTURES
Record Dates: First submitted 2022-08-19; First posted 2022-08-22 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Wound Heal
Keywords: wounds; superinfections; stitches
MeSH Terms: conditions — Wounds and Injuries; Superinfection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Identify the risk factors for complications as well as study the evolution of wounds sutured in the emergency room towards complications such as superinfections, necrosis, disunity of the stitches linked to inadequate initial care.

DETAILED DESCRIPTION:
All traumatic injuries should be considered contaminated upon presentation to the emergency room. This is why the main objective of this study was to describe the attitude of patients towards their wounds, to identify the risk factors for complications as well as to study the evolution of sutured wounds in the emergency room towards complications such as superinfections, necrosis, disunity of stitches linked to inadequate initial treatment.

This is a prospective, observational, monocentric study carried out in the emergency services of the Fattouma Bourguiba hospital in Monastir.

ELIGIBILITY:
Inclusion Criteria:

* Patients who presented to the ambulatory emergency circuit of the EPS Fattouma Bourguiba Monastir having as main reason for consultation an acute suturable wound.

Exclusion Criteria:

* Wounds requiring surgical treatment
* Septic wounds
* Chronic lesions
* Vascular wounds
* Patients who did not consent to the protocol.

Ages: 1 Year to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients with an acute suturable wound and accept to enroll the study .
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2022-08-08 (Actual); Primary Completion 2025-06-08 (Estimated); Study Completion 2025-10-10 (Estimated)

PRIMARY OUTCOMES:
Evolution of the wound and the healing period. | day 10
  After discharge from ED patients were called back in order to know information about the Suture complications(infection, release of stitches, hematoma, etc.)

CONTACTS AND LOCATIONS:
Overall Officials: Bel Haj Ali A Khaoula, MD, Study Director — CHU Fattouma Bourguiba Monastir, service des urgences
Locations (1):
- Nouira, Monastir, Tunisia

IPD SHARING:
Plan to Share IPD: No